CLINICAL TRIAL: NCT02085369
Title: Effect of Bariatric Surgery on Cognition, Genetics and Lifestyle
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PH2014; PH2014 (Other Grant/Funding Number: Uppsala University)
Record Dates: First submitted 2014-01-31; First posted 2014-03-12 (Estimated); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Obesity, Morbid
Keywords: Bariatric surgery; Cognitive function; Gene expression; Metabolomics; Obesity; Overweight; Lifestyle
MeSH Terms: conditions — Obesity, Morbid; Obesity; Overweight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A fasted blood sample (50 mL) will be taken before and 2h after a standardized meal.
  Through epigenetic study, we will analyze the changes in DNA methylation after surgery in genes related to metabolism (at the Science for Life Laboratory (SciLifeLab) with 450K Human Meth arrays).
  In addition, blood samples from these obese patients analyzed (before and after surgery) after ingestion of a predetermined test meal (for example, high protein) to explore changes in metabolites profile. Metabolites in the samples will be quantified by the SciLifeLab.
Oversight: Data Monitoring Committee: No

SUMMARY:
Obesity bariatric surgery patients usually lose more than 50% of their former obesity within a relatively short time (~ 2 years). There is still a lack of knowledge about underlying psychological and biological mechanisms of decline in body weight. The intention of this project is to investigate whether bariatric surgery is associated with patients' cognitive ability, lifestyle and/or gene expression and metabolomics.

ELIGIBILITY:
Inclusion Criteria:

* First bariatric surgery

Exclusion Criteria:

* More than one surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients with bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Changes in gene expression profile (a.o. FTO, BDNF) following a standardized meal (before vs. after surgery) | 1 year
  Gene expression profiling (whole genome analysis, with first interest in FTO and BDNF expression) to assess changes in gene expression before vs. after surgery, and to associate gene expression with weight loss after surgery

SECONDARY OUTCOMES:
The effect of bariatric surgery on cognitive functioning (inhibitory control, selective attention) | Measures 1 y, 2 y, and 5 y after surgery.
  No-Go go task (to assess inhibitory control) and Stroop tasks (to assess selective attention) will be measured to assess change in these cognitive functions before vs. after surgery, and to associate cognitive functioning with weight loss after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Magnus Sundbom, MD, Principal Investigator — Academic Hospital Uppsala; Helgi Schiöth, Prof, Study Director — Uppsala University; Olga Titova, PhD, Study Director — Uppsala University
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden